CLINICAL TRIAL: NCT04566224
Title: Comparison of Intubation Rate of Macintosh Size 2 and 3 Blades in Asian Female: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chun Lin, attending physician, department of anesthesiology, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11MMHIS107
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Intubation;Difficult
Keywords: Intubation rate; Macintosh blade; Asian women; intubation difficulty scale

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macintosh 2 group (Experimental): Using Macintosh size 2 blade for direct laryngoscope intubation according to randomization
  Interventions: Device: Macintosh size 2 blade
- Macintosh 3 group (Active Comparator): Using Macintosh size 3 blade for direct laryngoscope intubation according to randomization
  Interventions: Device: Macintosh size 3 blade

INTERVENTIONS:
Device: Macintosh size 2 blade — intubate with Macintosh size 2 blade
  Arms: Macintosh 2 group
Device: Macintosh size 3 blade — intubate with Macintosh size 3 blade
  Arms: Macintosh 3 group

SUMMARY:
Direct laryngoscope is a standard equipment for endotracheal intubation. To identify the differences between Macintosh size 3 and 2 blades, we will analysis the data collected from airway and intubation condition.

DETAILED DESCRIPTION:
Selection the most appropriate size of laryngoscope blade size could not only increased intubation successful rate at the first time but also decrease the incidence of tissue trauma. Laryngoscope blade used in daily practice is usually Macintosh 3. However, compared with Caucasian people, Asian people are smaller and thinner especially in women. This study aims to confirm that the Macintosh 2 blade is not inferior to size 3 blade in laryngeal view and intubation rate.

Female patients without known difficult airway will be enrolled and allocated into Macintosh blade size 2 and size 3 groups. The age, body weight, body height, Mallampati classification, mouth opening, thyromental distance, neck circumference, intubation time, Cormack-Lehane grade, intubation difficulty scale scores and associated teeth or tissue traumas will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* with American Society of Anesthesiologists (ASA) physical status classification 1, 2, or 3
* undergo elective surgery
* receive endotracheal intubation

Exclusion Criteria:

* with known difficult airway (i.e. pathology of the neck, upper airway or alimentary tracts)
* with risks of pulmonary aspiration (i.e. emergent operation, pregnancy or inadequate nil per os)
* with previous difficult intubation history
* intubation attempts more than three times
* patient refusal

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2012-05-31 (Actual)

PRIMARY OUTCOMES:
Intubation time | 0-10 minutes during induction
  Time from laryngoscope insertion to the first adequate lung insufflation
Cormack-Lehane grade | 0-10 minutes during induction
  Classification of glottis view during intubation
Intubation difficulty scale scores | 0-10 minutes during induction
  Scoring system to assess the difficulty of intubation in each patient
Tissue trauma | 0-10 minutes during induction
  Any tissue trauma event related to intubation
Teeth trauma | 0-10 minutes during induction
  Any dental damage event related to intubation

CONTACTS AND LOCATIONS:
Overall Officials: Nuan-Yen Su, MS, Study Director — Mackay Memorial hospital, department of anesthesiology, attending physician
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellick LB, Edholm T, Corbett SW. Pediatric laryngoscope blade size selection using facial landmarks. Pediatr Emerg Care. 2006 Apr;22(4):226-9. doi: 10.1097/01.pec.0000210171.17892.7a. PMID 16651910
- [Background] Ashfaque M, Mason J, Al-Shaikh B, Adegoke K. A comparison of the Laryngopharyngeal Examination blade and the English Macintosh laryngoscope blade using an intubating manikin: a prospective randomized crossover study. Eur J Anaesthesiol. 2009 Nov;26(11):917-22. doi: 10.1097/EJA.0b013e32832c7848. PMID 19593148
- [Background] Asai T, Matsumoto S, Fujise K, Johmura S, Shingu K. Comparison of two Macintosh laryngoscope blades in 300 patients. Br J Anaesth. 2003 Apr;90(4):457-60. doi: 10.1093/bja/aeg086. PMID 12644417
- [Background] Watanabe S, Suga A, Asakura N, Takeshima R, Kimura T, Taguchi N, Kumagai M. Determination of the distance between the laryngoscope blade and the upper incisors during direct laryngoscopy: comparisons of a curved, an angulated straight, and two straight blades. Anesth Analg. 1994 Oct;79(4):638-41. doi: 10.1213/00000539-199410000-00004. PMID 7943768